CLINICAL TRIAL: NCT01960868
Title: Early Rehabilitation Program is Feasible and Safe in ICU in Liver Transplanted Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A00760-45; 2013-20 (Other: AP HM)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Liver Transplanted Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients (Experimental)
  Interventions: Other: experimental physical therapy
- control group (Other)
  Interventions: Other: standard physiotherapy

INTERVENTIONS:
Other: standard physiotherapy
  Arms: control group
Other: experimental physical therapy
  Arms: patients

SUMMARY:
Liver transplantation is the last surgical treatment for patients with acute or chronic liver disease. Transplantation therapies technics are in constant evolution. It allows an increasing survivals rates and time to come back to daily activities. The postoperative treatment after abdominal surgery as Liver Transplantation (LT) is usually performed in Intensive Care Unit (ICU).This postoperative phase is one of the most important steps regarding the involvement of the rehabilitation of the patient (Rongies 2005). Physical abilities transplantation are likely to be important in the postoperative. It appears that pre-transplant subjects have a weakened muscle potential, they will increase it significantly in the months after transplantation with a rehabilitation program adapted (Beyer 1999). Length of stay in ICU depends on surgery complications. Inactivity induced by sedation and ICU length of stay are major factor for increasing complications as respiratory disorders and muscle weakness. Several studies have reported feasibility and safety an early mobility program in ICU, especially regarding the length of stay decrease (Bailey 2007; Morris 2008; Schweickret 2009, Needham 2010; Bourdin 2010) These early mobility programs encompass muscle strength assessment, passive range of motion, active mobility, sitting on the edge of bed, standing and walking, which would be related to the primary disease of LT (Rongies 2008). The assessment of the strength for ICU patient is feasible and reproducible with the Medical Research Council score (MRC score). The MRC score consists in an assessment of three muscle groups of upper and lower limbs. Sitting positions and verticalization are included in programs begun as soon as possible after surgery evaluation of the response level to verbal stimulation and physical abilities (Gosselink 2011). The skills of the physiotherapist are established in legal texts making him a key in the assessment and management of these patients on musculoskeletal and respiratory domains.

The purpose of this study is to validate data feasibility and tolerance. Another aim is also to assess the length of stay in ICU, of early mobility and physical program, started in the postoperative period in a population of patients with liver transplantation, during their stay in ICU of Prof. Albanese. Thus, we decided to carry out a parallel study, open, randomized monocentric comparing two groups of patient liver transplanted. The control group will receive the standard treatment used in the ICU and the experimental group will receive a protocol of early mobilization according to data from recent literature on the subject. The study is scheduled to last over one year and included patients will receive physical therapy on five days a week with a frequency of one to several times per day depending on the clinical requirements or conditions of the study.

ELIGIBILITY:
Inclusion Criteria:

* patient more than 18 years,
* patient for a liver transplant
* patient that informed consent was obtained

Exclusion Criteria:

* patient whose consent has not been obtained,
* patient with major cons-indications to the application program (paralysis neuromyopathy majeure),
* patient with hemodynamic instability or severe infection,
* pregnant women,
* nursing mothers,
* persons deprived of their liberty by a judicial or administrative decision,
* patient being a measure of legal protection,
* patient requiring a transplant urgently
* patient younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Medical Research Council score (MRC score). | 12 months
  The assessment of the strength for ICU patient

SECONDARY OUTCOMES:
the length of stay in ICU, | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Maffei P, Wiramus S, Bensoussan L, Bienvenu L, Haddad E, Morange S, Fathallah M, Hardwigsen J, Viton JM, Le Treut YP, Albanese J, Gregoire E. Intensive Early Rehabilitation in the Intensive Care Unit for Liver Transplant Recipients: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1518-1525. doi: 10.1016/j.apmr.2017.01.028. Epub 2017 Mar 6. PMID 28279659